CLINICAL TRIAL: NCT02975154
Title: Microcurrent Therapy in the Treatment of Osteoarthritis of the Knee: a Randomized, Controlled Pilot Study
Brief Title: Microcurrent Therapy in the Treatment of Osteoarthritis of the Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Federal Ministry for Economic Affairs and Energy (Other)
Responsible Party: Principal Investigator, PD Dr. Martin Weigl, MPH, PD, MD, MPH (Harvard University), Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MicrocurrencyOA
Record Dates: First submitted 2016-11-21; First posted 2016-11-29 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Osteoarthritis,Knee
Keywords: osteoarthritis; microcurrent; knee; electrotherapy
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Microcurrent therapy, type A (Active Comparator): Microcurrent therapy: Channel A: 100 µA; 200 Hz; Channel B: 100 µA; 300 Hz. Duration of each treatment session: 30 minutes. Number of sessions: 10.
  Previous treatments will be continued.
  Interventions: Device: Microcurrent therapy
- Microcurrent therapy, type B (Active Comparator): Microcurrent therapy: Channel A: 25 µA; 200 Hz; Channel B: 100 µA; 300 Hz. Duration of each treatment session: 30 minutes. Number of sessions: 10. Previous treatments will be continued.
  Interventions: Device: Microcurrent therapy
- Sham Microcurrent therapy (Sham Comparator): Microcurrent therapy: Channel A: 0 µA; 0 Hz; Channel B: 0 µA; 0 Hz. Duration of each treatment session: 30 minutes. Number of sessions: 10. Previous treatments will be continued.
  Interventions: Device: Microcurrent therapy
- No Intervention (No Intervention): No Intervention. Previous treatments will be continued.

INTERVENTIONS:
Device: Microcurrent therapy — The microcurrent therapy will be applied with electrodes that are fixed around the knee. The two electrodes of channel A will be placed at the inner and outer side of the knee that is most affected by pain. The two electrodes of channel B will be placed above and below the patella. An apparatus with CE certificate will be used.
  Arms: Microcurrent therapy, type A; Microcurrent therapy, type B; Sham Microcurrent therapy

SUMMARY:
This study evaluates the effect of Microcurrent Therapy in the treatment of osteoarthritis of the knee. Patients will be randomized to four groups: Group 1 and 2 both will receive Microcurrent Therapy, but different currents will be used. Group 3 will receive treatment with the Microcurrent treatment apparatus, but without any current. Group 4 will be a control group without specific interventions.

DETAILED DESCRIPTION:
The objective of this randomized, controlled pilot study is to evaluate the effect of Microcurrent therapy on pain and physical function in patients with osteoarthritis of the knee. The secondary objective is to compare the effects of different currents. Patients will be randomized to four groups: Group 1 and 2 both will receive Microcurrent Therapy, but different currents will be used. Group 3 will receive treatment with the Microcurrent treatment apparatus, but without any current. Group 4 will be a control group without specific intervention.

Group 1, 2 and 3 will receive 10 sessions of treatment in a treatment phase of four weeks. Assessments for group 1, 2, and 3 will be scheduled for screening (T0), at the first day of treatment (T1), at the end of treatment (T2) and three months after the end of treatment (T3). Group 4 will be assessed at a screening visit T0, at T1, at T2 (approximately 21 days after T1), and at T3 (three months after T2). Patients will be recruited based on the records of the clinic.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis of the knee
* pain intensity > 3 on the numerical rating scale (0-10)

Exclusion Criteria:

* knee arthroplasty
* gravity
* dermal Irritation at the skin of the knee
* carcinoma
* known osteoarthritis grade 4 (Kellgren and Lawrence score)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2017-09-04 (Actual); Study Completion 2017-09-04 (Actual)

PRIMARY OUTCOMES:
Numerical Ratings scale (NRS) for pain (0-10) | Change of NRS: Before treatment vs. end of treatment (in average 21 days later)
  numerical Rating scale

SECONDARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score | Change of scores: Before treatment vs. end of treatment (in average 21 days later)
  Knee specific Instrument measuring pan, function and Quality of life.
Short-Form 36 | Change of scores: Before treatment vs. end of treatment (in average 21 days later)
  Generic HRQOL measure
Satisfaction with Treatment (Questionnaire) | Evaluation at the end of treatment (in average 21 days after Start of treatment)
  Self-administered questionnaire that was developed for this study
Range of Motion knee joint | Change: Before treatment vs. end of treatment (in average 21 days later)
  Clinical test with goniometer
Get-up-and-Go-Test (GUG) | Change: Before treatment vs. end of treatment (in average 21 days later)
  clinical test that measures mobility
6-minute walking test | Change: Before treatment vs. end of treatment (in average 21 days later)
  Clinical test that measures the Walking ability

CONTACTS AND LOCATIONS:
Overall Officials: Martin B Weigl, Principal Investigator — Department of Orthopedics, Physical Medicine and Rehabilitation, University Hospital Munich, Ludwig Maximilians University Munich
Locations (1):
- Ludwig Maximilian University, University Hosipital, Department of Orthopedics, Physical Medicine and Rehabilitation, Munich, Germany

IPD SHARING:
Plan to Share IPD: No